CLINICAL TRIAL: NCT01038700
Title: Impact du Vieillissement (VI) Sur le Compartiment Circulant et Sur la Mobilisation (MO) Des progéniteurs endothéliaux (PE) Par ischémie Locale (IL) : étude Pilote
Brief Title: Circulating Endothelial Compartment During Normal and Pathological Aging
Acronym: VIMOPEIL
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation pour la Recherche Médicale (Other); Assistance Publique Hopitaux De Marseille (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Yannick VACHER, Department Clinical Research of devloppement
Other Study IDs: P070801
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Circulating endothelial compartment; microparticles; endothelial progenitors cells; circulating endothelial cells; transcriptome; aging; Healthy volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This part of the project aims to describe changes in markers of vascular competence (Endothelial Microparticles Platelet (EMP), Circulating endothelial cells (CEC) and Circulating endothelial progenitors (EPC)) at different ages of lifespan both in physiological state and in response to hypoxia-induced vascular stress.

DETAILED DESCRIPTION:
Blood will be harvested in citrated or EDTA anticoagulant and processed within one hour for Endothelial Microparticles Platelet (EMP), Circulating endothelial cells (CEC) and Circulating endothelial progenitors (EPC) determination.

Methods for endothelial marker determination:

* Endothelial Microparticles Platelet free plasma (PFP) will be prepared by a double step centrifugation of citrated blood at 1,500g for 15 min and 13,000 g for 2 min at room temperature. Then EMP will be enumerated by flow cytometry after labelling of PFP using monoclonal antibodies directed against endothelial antigens, such as CD144 (19). To investigate the proportion of EMP within the whole circulating MP, MP for platelet, leukocyte and erythrocyte origins will be determined using respectively, CD41, CD45, Glycophorin-directed antibodies, and the total number of phosphatidylserine expressing MP will be determined using AnnexinV binding.
* CEC will be enumerated using the consensual methodology based on an immunomagnetic separation assay (20). CEC will be isolated from EDTA whole blood using magnetic beads coated with antibodies directed against the CD146 antigen. Isolated cells will be identify using additional criteria such as morphology, size higher than 15µm, cell rosettes bearing more than 5 beads, and expression of endothelial markers (lectin binding).
* For EPC two complementary approaches will be used for determination:

  1. Flow cytometry after direct immunolabelling of whole blood or the mononuclear cell fraction using monoclonal antibodies and viability marker 7AAD. Due to the lack of specific markers for EPC and the great heterogeneity of cells that recovered the features of EPC21 flow cytometry analysis will include the numeration of different cell populations corresponding to differentiation state of EPC: CD34+CD133+ cells and CD34+KDR+ cells. The circulating haematopoietic progenitors CD34+CD45+ will be also numbered.-
  2. Clonogenic assays allowing the numeration of Colony Forming Unit after ex vivo culture of EPC including: - CFU-EC, which are EPC of myeloid subtype (also called early EPC) will be determined according to the previously described method of Hill et al. The non-adherent fraction of mononuclear cells will be plated on fibronectin coated dishes in Endocult® medium. the number of endothelial colonies will be counted after a 48h culture - High Proliferative Potential CFU, which are true angioblasts will be determined by Ingram's method (21). Mononuclear cells are plated on fibronectin-coated plates in EGM-2MV culture medium and late EPC colonies are enumerated after 10-15 days of culture. - three-dimension methyl cellulose assay in which the only added growth factor is VEGF. The CFU-EC are numbered after 14 days as usually performed for haematopoietic stem cells. Effect of hypoxia on the equilibrium between endothelial damage and repair According to Ingram, the normal vascular endothelium contains high proliferating potency EPC (22) suggesting that late EPC may also originate from the vessel wall. In addition, local hypoxia might also mobilize EPC (23).

We designed a protocol which specific aims are 1/ to test the effect of local hypoxia on the markers of endothelial damage/repair equilibrium 2/ to define whether in elderly patients, local ischemia can be used to mobilize EPC and to increase their proliferation potential compared to EPC isolated in resting conditions. Two groups of healthy volunteers aged 20-30 and 60-70 years from our cohorts will be submitted to forearm transient ischemia as described by Friedrich et al (23). Peripheral blood samples will be obtained before and after 10 min of venous occlusion performed with a cuff pressure midway between systolic and diastolic pressure (24). EPC, CEC and EMP will be enumerated according to the methods described supra and EPC will be tested for proliferating capacity at each time point. The arterial phenotype of conducting arteries will be evaluated, by the acute flow-mediated vasodilatation (FMD) and endothelium-independent vasodilatation (EIV) of the brachial artery (BA) in young and older healthy volunteers using a high-resolution echotracking system. The efficiency of venous occlusion will be evaluated by the release of t-PA by endothelial cells.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of 20-30 and 60-70 years old
* Non smokers male
* Biological test in normal values : lipids, glucose, TGO, TGT, alkaline phosphatases, gamma-GT, bilirubin, creatinine, ionogram, Ca++, albumin, proteins, WBC, platelets count, coagulation tests (APTT, PT, Fibrinogen).
* Negative HIV1 and 2, HBV (Hbs antigen) and HCV serology.
* Normal ECG 12 derivations, arterial pressure and cardiac frequency.

Exclusion Criteria:

* Evaluative disease in the past 10 days
* Hemorrhagic disorders
* Treatments with antiplatelets agents, oral or injectable anticoagulant
* Statins, glitazones, EPO, G-CSF
* Frequent faintness
* Blood donation in the 3 months preceding the study
* People in period of exclusion on the National File of the people who lend themselves to biomedical research
* Refusal or linguistic or psychic incapacity to sign the enlightened consent
* Biological parameters apart from the usual values of the healthy subject (Hb<10 g/dL, TGO/TGT > 2 times higher limit of normal values)
* Prone not being able to subject to the constraints protocol (for example, not cooperating, incompetent to go to the visits of follow-up and probably incompetent to finish the study).

Ages: 10 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2008-12; Primary Completion 2009-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Analyse of CEC, EMP and EPC at different ages of lifespan both in physiological state and in response to an hypoxia- induced vascular stress | 3 days

SECONDARY OUTCOMES:
Transcriptome analysis on EPC isolated from cord blood and peripheral blood from young and old adults | end

CONTACTS AND LOCATIONS:
Overall Officials: David SMADJA, PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hegp- Cic, Paris, France

REFERENCES:
- [Derived] HoWangYin KY, Loinard C, Bakker W, Guerin CL, Vilar J, d'Audigier C, Mauge L, Bruneval P, Emmerich J, Levy BI, Pouyssegur J, Smadja DM, Silvestre JS. HIF-prolyl hydroxylase 2 inhibition enhances the efficiency of mesenchymal stem cell-based therapies for the treatment of critical limb ischemia. Stem Cells. 2014 Jan;32(1):231-43. doi: 10.1002/stem.1540. PMID 24105925
- [Derived] Evrard SM, d'Audigier C, Mauge L, Israel-Biet D, Guerin CL, Bieche I, Kovacic JC, Fischer AM, Gaussem P, Smadja DM. The profibrotic cytokine transforming growth factor-beta1 increases endothelial progenitor cell angiogenic properties. J Thromb Haemost. 2012 Apr;10(4):670-9. doi: 10.1111/j.1538-7836.2012.04644.x. PMID 22284809